CLINICAL TRIAL: NCT05609344
Title: Barbershop Talk: Reducing Excessive Alcohol Consumption Among Men
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Health Services Research
Other Study IDs: 273439
Record Dates: First submitted 2022-10-17; First posted 2022-11-08 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-04

CONDITIONS: Drinking Behavior; Drinking Excessive; Drinking
MeSH Terms: conditions — Drinking Behavior

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SBIRT (Experimental): Each intervention barbershop, will hold screening days, where a trained community health worker will be onsite to provide Screening, Brief Intervention, and Referral to Treatment (SBIRT).
  Interventions: Behavioral: SBIRT
- Usual-care (Other): Six months after completion of Time 1, barbershops in the usual-care arm will receive the intervention.
  Interventions: Behavioral: SBIRT

INTERVENTIONS:
Behavioral: SBIRT — Low risk individuals will receive an educational pamphlet about alcohol use and the impact on health. Moderate Risk individuals will receive a brief alcohol intervention. High risk individuals will receive the brief alcohol intervention and be referred to specialty treatment.

SUMMARY:
Unhealthy drinking is considered one of the top 10 public health concerns in the United States. Not only has heavy drinking been linked to poorer overall health and the chances of getting cancer and cardiovascular diseases, but it also causes about 88,000 deaths and 2.5 million years of potential life lost each year in the U.S. Men living in rural areas tend to drink more. In Arkansas, a rural state with high rates of unhealthy drinking, men are more likely to report heavy drinking (4 or more drinks a day) and to drink more when binge drinking. Screening, Brief Intervention, and Referral to Treatment (SBIRT) is an evidence-based, multilevel, integrated public health approach for early intervention and timely referral to more intensive treatment for those with substance use disorders. SBIRTs have been successfully used in primary care and emergency settings.

However, men in rural areas may lack access to evidence-based care for unhealthy drinking due to many factors, including limited healthcare providers and insurance standing. Given the increased chances of death and illness linked to harmful drinking among rural men and the serious health consequences involved, it is urgent to improve access to evidence-based care. This can be achieved by expanding services into community settings that men in rural areas are more likely to visit, such as barbershops. Thus, the goals of this proposed Hybrid Type 2 pragmatic effectiveness-implementation trial are to: 1) test the effectiveness of an evidence-based SBIRT intervention for use within barbershops (Barbershop Talk); and 2) generate the scientific evidence needed to implement SBIRTs in "real world" settings. Data from this study will further our understanding of how to reduce the chances of experiencing alcohol attributable morbidity and mortality among men living in rural areas. Data will also enhance our understanding of strategies that can improve the implementation of evidence-based care models in non-clinical settings, thereby extending the reach of evidence-based care to rural communities with high needs.

ELIGIBILITY:
Inclusion Criteria:

* male
* aged 18 or older
* resident of Arkansas

Exclusion Criteria:

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 600 (Estimated)
Dates: Start 2023-06-26 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Alcohol Use - total number of drinking days | Baseline
  At-risk drinking behavior measured as:
  number of drinking days
Alcohol Use - total number of drinking days | 3 months
  At-risk drinking behavior measured as:
  number of drinking days
Alcohol Use - total number of drinking days | 6 months
  At-risk drinking behavior measured as:
  number of drinking days
Alcohol Use - number of unhealthy drinking days | Baseline
  At-risk drinking behavior measured as:
  number of unhealthy drinking days
Alcohol Use - number of unhealthy drinking days | 3 months
  At-risk drinking behavior measured as:
  number of unhealthy drinking days
Alcohol Use - total number of unhealthy drinking days | 6 months
  At-risk drinking behavior measured as:
  number of unhealthy drinking days
Mental Health - depression | Baseline
  The PHQ-9 is the depression module of the Patient Health Questionnaire (a diagnostic instrument for common mental disorders), which scores each of the 9 DSM-IV criteria as "0" (not at all) to "3" (nearly every day). The PHQ9 will be used for this outcome.
Mental Health - depression | 3 months
  The PHQ-9 is the depression module of the Patient Health Questionnaire (a diagnostic instrument for common mental disorders), which scores each of the 9 DSM-IV criteria as "0" (not at all) to "3" (nearly every day). The PHQ9 will be used for this outcome.
Mental Health - depression | 6 months
  The PHQ-9 is the depression module of the Patient Health Questionnaire (a diagnostic instrument for common mental disorders), which scores each of the 9 DSM-IV criteria as "0" (not at all) to "3" (nearly every day). The PHQ9 will be used for this outcome.
Mental Health - Posttraumatic Stress Disorder (PTSD) | Baseline
  Posttraumatic Stress Disorder Checklist for DSM-5 (PCL5)
Mental Health - Posttraumatic Stress Disorder (PTSD) | 3 months
  Posttraumatic Stress Disorder Checklist for DSM-5 (PCL5)
Mental Health - Posttraumatic Stress Disorder (PTSD) | 6 months
  Posttraumatic Stress Disorder Checklist for DSM-5 (PCL5)
Social Support | Baseline
  Family, friend, and partner support (number of people in support network)
Social Support | 3 months
  Family, friend, and partner support (number of people in support network)
Social Support | 6 months
  Family, friend, and partner support (number of people in support network)
Healthcare Utilization | Baseline
  Number of subjects who have utilized healthcare services
Healthcare Utilization | 3 months
  Number of subjects who have utilized healthcare services
Healthcare Utilization | 6 months
  Number of subjects who have utilized healthcare services

CONTACTS AND LOCATIONS:
Overall Officials: Tiffany F Haynes, PhD, Principal Investigator — University of Arkansas
Locations (1):
- UAMS, Little Rock, Arkansas, United States